CLINICAL TRIAL: NCT05411991
Title: Diuretic Treatment in Acute Heart Failure With Volume Overload Guided by Serial Spot Urine Sodium Assessment
Acronym: DECONGEST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Roche Diagnostics GmbH (Industry); Jessa Hospital (Other)
Responsible Party: Principal Investigator, Frederik Hendrik Verbrugge, MD PhD MSc, Head of Clinic/Assistant Professor, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC-2021-236; 2021-005426-18 (EudraCT Number)
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Acute Heart Failure; Diuretics Drug Reactions
Keywords: Acute Heart Failure; Natriuresis; Diuretics; Edema
MeSH Terms: conditions — Edema | interventions — Acetazolamide; Bumetanide; Chlorthalidone; Canrenoic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): Application of a standardized diuretic schedule with following key components:
  * UNa assessment in spot urine sample after every bolus of loop diuretics with continuation of intravenous diuretics until absence of clinical signs of fluid overload AND UNa <80 mmol/L
  * Loop diuretic dosing according to estimated glomerular filtration rate (eGFR) with higher dose for lower eGFR
  * Upfront use of intravenous acetazolamide 500 mg OD unless hypernatremia or metabolic acidosis
  * Upfront use of oral chlorthalidone 50 mg OD if eGFR <30 mL/min/1.73m² OR hypernatremia
  * Full nephron blockade with intravenous acetazolamide 500 mg OD, intravenous bumetanide 4 mg TID, oral chlorthalidone 100 mg OD, and intravenous canrenoate 200 mg OD in case of diuretic resistance, defined as UNa <80 mmol/L and persistent clinical signs of fluid overload
  * Provision of 500 mL intravenous Dextrose 5% with 3 g MgSO4 and 40 mmol KCl daily during intravenous diuretics
  Interventions: Diagnostic Test: UNa measurement after intravenous loop diuretic bolus; Drug: Intravenous acetazolamide 500 mg OD; Drug: Intravenous bumetanide TID; Drug: Oral chlorthalidone OD; Drug: Intravenous canrenoate 200 mg OD; Other: Maintenance infusion; Drug: Oral potassium supplements; Other: Intravenous hypertonic saline; Other: Switch to oral diuretic therapy
- Control arm (Active Comparator): Usual care for AHF. It is recommended to administer an intravenous loop diuretic dose at least BID (or through continuous infusion), with the aim of achieving a urine output 3-5 L per day until the patient is considered in an optimal volume status as is recommended by current guidelines. Urine electrolyte assessment in the control arm is not allowed as it is a key component of the studied intervention.
  Interventions: Other: Usual AHF care

INTERVENTIONS:
Diagnostic Test: UNa measurement after intravenous loop diuretic bolus — Sodium concentration is measured on a urine spot sample, collected 30-120 min after administration of every protocol-specified intravenous bumetanide dose.
  Arms: Intervention arm
Drug: Intravenous acetazolamide 500 mg OD — Upfront use of intravenous acetazolamide 500 mg OD as part of the diuretic treatment, unless hypernatremia (>145 mmol/L) or metabolic acidosis (bicarbonate <22 mmol/L) is present at the moment of the scheduled administration.
  Other Names: Diamox (brand name for acetazolamide)
  Arms: Intervention arm
Drug: Intravenous bumetanide TID — An intravenous bolus of bumetanide is administered TID, with dosing according to eGFR: 2 mg for an eGFR >45 mL/min/1.73m²; 3 mg for an eGFR 30-45 mL/min/1.73m²; and 4 mg for an eGFR <30 mL/min/1.73m². At any time diuretic resistance is encountered (persistent clinical signs of fluid overload with UNa <80 mmol/L), a dose of 4 mg TID is used.
  Other Names: Burinex (brand name for bumetanide)
  Arms: Intervention arm
Drug: Oral chlorthalidone OD — In case of hypernatremia (>145 mmol/L) or low eGFR (<30 mL/min/1.73m²), oral chlorthalidone 50 mg OD is added to the diuretic treatment. At any time diuretic resistance is encountered (persistent clinical signs of fluid overload with UNa <80 mmol/L), oral chlorthalidone is provided at a dose of 100 mg OD. Chlorthalidone is never administered in case of hypotonic hyponatremia with serum sodium concentration <135 mmol/L.
  Other Names: Hygroton (brand name for chlorthalidone)
  Arms: Intervention arm
Drug: Intravenous canrenoate 200 mg OD — At any time diuretic resistance is encountered (persistent clinical signs of fluid overload with UNa <80 mmol/L), intravenous canrenoate 200 mg OD is provided. Canrenoate is never administered in case of hypotonic hyponatremia with serum sodium concentration <135 mmol/L or if serum potassium levels are >5.5 mmol/L. If canrenoate is administered, oral mineralocorticoid receptor drugs are temporarily withhold until switch to oral diuretic treatment.
  Other Names: Soldactone (brand name for canrenoate)
  Arms: Intervention arm
Other: Maintenance infusion — A maintenance infusion with 500 mL dextrose 5% and 3 g MgSO4 is started at an infusion rate of 20 mL/h upon the moment of first protocol-specified administration of intravenous diuretics and continued until switch to oral diuretic therapy. 40 mmol KCl is added if serum potassium levels are <4 mmol/L. In case of hypotonic hyponatremia with serum sodium concentration <130 mmol/L, dextrose 5% will not be provided and MgSO4 will be administered in 50 mL of normal saline (NaCl 0.9%).
  Arms: Intervention arm
Drug: Oral potassium supplements — If serum potassium levels are <3.5 mmol/L at any time during the administration of intravenous diuretics, oral potassium supplements are provided as needed to keep serum potassium levels >4 mmol/L
  Other Names: KCl
  Arms: Intervention arm
Other: Intravenous hypertonic saline — In case of hypotonic hyponatremia with serum sodium concentration <125 mmol/L, a bolus of 150 mL hypertonic saline 3% is administered and repeated OD if necessary, until sodium levels are ≥135 mmol/L.
  Arms: Intervention arm
Other: Switch to oral diuretic therapy — Upon complete resolution of clinical signs of fluid overload with UNa <80 mmol/L, intravenous diuretics are switched to an oral schedule including:
  * Loop diuretics with dose & frequency at the discretion of the treating physician
  * Chlorthalidone 50 mg if added for diuretic resistance at any time during the intravenous diuretic phase
  * Spironolactone 25 mg or another equivalent mineralocorticoid receptor antagonist
  Arms: Intervention arm
Other: Usual AHF care — It is recommended to administer an intravenous loop diuretic dose at least BID (or through continuous infusion), with the aim of achieving a urine output 3-5 L per day until the patient is considered in an optimal volume status as is recommended by current guidelines.
  Arms: Control arm

SUMMARY:
This is a pragmatic, multicenter, interventional, parallel-arm, randomized, open-label trial to investigate whether a diuretic regimen, based on serial assessment of sodium concentration (UNa) on spot urine samples after diuretic administration and with low-threshold use of combination diuretic therapy, improves decongestion versus usual care in acute heart failure (AHF), potentially leading to better clinical outcomes.

DETAILED DESCRIPTION:
Key interventions are:

* Assessment of UNa in spot urine samples after every bolus administration of loop diuretics with continuation of intravenous diuretics until resolution of clinical signs of fluid overload AND UNa <80 mmol/L
* Dosing of loop diuretic bolus according to estimated glomerular filtration rate (eGFR)
* Upfront use of intravenous acetazolamide 500 mg OD unless hypernatremia (>145 mmol/L) or metabolic acidosis (bicarbonate <22 mmol/L)
* Upfront use of oral chlorthalidone 50 mg OD if eGFR <30 mL/min/1.73m² OR hypernatremia (>145 mmol/L)
* Switch to full nephron blockade with intravenous acetazolamide 500 mg OD, intravenous bumetanide 4 mg TID, oral chlorthalidone 100 mg OD, and intravenous canrenoate 200 mg OD in case of diuretic resistance, defined as UNa <80 mmol/L and persistent clinical signs of fluid overload
* Provision of 500 mL intravenous Dextrose 5% with 3 g MgSO4 and 40 mmol KCl daily during diuretic therapy with intravenous diuretics

ELIGIBILITY:
Inclusion criteria:

* At least 18 y/o and able to provide informed consent
* Hospital admission (anticipated stay >24 h after randomisation) with diagnosis of acute heart failure according to the treating physician
* At least one of the following three signs of volume overload:

  1. bilateral oedema 2+, indicating clear pitting
  2. ascites that is amenable for drainage, confirmed by echography (no obligation to perform abdominal echocardiography, but necessary when presence of ascites is used as an entry criterion for the study)
  3. uni- or bilateral pleural effusions that are amenable for drainage, confirmed by chest X-ray or lung ultrasound (no obligation to perform chest X-ray, but necessary when presence of pleural effusions is used as an entry criterion for the study)
* Plasma NTproBNP level >1,000 ng/L

Exclusion criteria:

* No possibility to collect reliable urine spot samples after diuretic administration
* Administration of any diuretic within 6 h before randomisation, except for a mineralocorticoid receptor antagonist or sodium glucose co-transporter-2 inhibitor as part of the patient's maintenance treatment for heart failure. Patients can still be included after withholding these diuretics for 6 h, after which randomisation can be performed if they qualify all other criteria.
* Severe kidney dysfunction, defined as an eGFR <15 mL/min/1.73m² calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula and/or previous, current, or planned future renal replacement therapy
* Systolic blood pressure <90 mmHg, mean arterial pressure <65 mmHg, or need for inotropes/vasopressor therapy at randomisation
* Any acute coronary syndrome within 30 days prior to enrolment, defined as typical chest pain with a troponin rise above the 99th percentile of normal and/or electrocardiographic changes suggestive of cardiac ischemia
* History of heart or kidney transplantation
* History of mechanical circulatory support
* Known obstructive hypertrophic cardiomyopathy, congenital heart disease, acute mechanical cause of acute heart failure (e.g., papillary muscular rupture), acute myocarditis, or constrictive pericarditis according to the treating physician
* Pregnant or breastfeeding woman
* Concomitant participation in another interventional study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2022-06-12 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederik H Verbrugge, M.D.; Ph.D.; M.Sc., Principal Investigator — Vrije Universiteit Brussel
Locations (2):
- Belgium (2):
  - University Hospital Brussels, Jette, Brussels Capital
  - Jessa Hospital, Hasselt, Limburg

IPD SHARING:
Plan to Share IPD: Yes
IPD will be made available upon reasonable request in adherence with transparency conventions in medical research and through requests to the chief investigator (Frederik H. Verbrugge, frederik.verbrugge@uzbrussel.be). The executive committee of DECONGEST has developed a comprehensive analysis plan and numerous prespecified analyses, which will be presented in future scientific presentations and publications. At a later time point, the full database will be made available in adherence with the ratified transparency policy.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol will be shared through clinicaltrials.gov immediately upon release. The statistical analysis plan will be shared before database lock at the end of the study.

REFERENCES:
- [Background] Vanhentenrijk S, Verbeeck J, Kalpakos T, Vandoren V, Braeckeveldt L, L'hoyes W, Choustoulakis E, Roosens B, Tang WHW, Verwerft J, Verbrugge FH. Rationale and Design of the DECONGEST (Diuretic Treatment in Acute Heart Failure With Volume Overload Guided by Serial Spot Urine Sodium Assessment) Study. J Card Fail. 2025 Apr;31(4):651-660. doi: 10.1016/j.cardfail.2024.08.044. Epub 2024 Aug 30. PMID 39218247

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Arm: Application of a standardized diuretic schedule with following key components:
  * Serial post-diuretic spot urine sodium (UNa) assessment
  * Loop diuretic dosing according to estimated glomerular filtration rate (eGFR)
  * Upfront use of intravenous acetazolamide 500 mg OD
  * Upfront use of oral chlorthalidone 50 mg OD if eGFR <30 mL/min/1.73m² OR hypernatremia
  * Full nephron blockade for diuretic resistance
  * Provision of 500 mL intravenous Dextrose 5% with 3 g MgSO4 and 40 mmol KCl daily during intravenous diuretics
Period: Overall Study
Arm/Group | Intervention Arm | Control Arm
Started | 53 | 54
Completed | 52 | 51
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Control Arm | Total
Number analyzed (Participants) | 52 | 51 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 81 (10) | 79 (10) | 80 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 45
  Male | 31 | 27 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 49 | 49 | 98
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
NTproBNP (ng/L) [Median (Inter-Quartile Range); unit: ng/L] | 4134 [2423 to 7920] | 4989 [2523 to 9014] | 4622 [2491 to 8824]

OUTCOME MEASURES:

1. Primary Outcome: Mortality, Days in Hospital & Decongestion
Description: The net treatment benefit is calculated for the hierarchical composite primary endpoint. Every patient from the intervention group is pair-wise compared with each patient from the control group to declare a winner or tie. The following criteria are sequentially assessed to declare a winner or a tie:
  1. Any subject surviving until 30 days after randomization wins from a subject who died. If both subjects did not survive until day 30, there is a tie.
  2. In a pair of subjects, both surviving up till day 30, the subject with the highest number of days alive and out of hospital or care facility during the 30-day follow-up window is declared the winner.
  3. In a pair of subjects, both surviving up till day 30 with the same number of days alive and out of hospital/care facility, the subject with the greatest relative reduction in NTproBNP from baseline is the winner (rounded to the closest percentage with a minimal difference of 5%). If the difference is <5%, there is a tie.
Time Frame: 30 days
Measure: Number; unit: % wins
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 52 | 51
% wins | 54.68 | 44.16
Statistical Analysis 1: Comparison: Intervention Arm vs Control Arm; Test type: Superiority; p = 0.357, General pairwaise comparison; Net treatment benefit = 10.5, 95% CI 2-sided [-11.9 to 31.9]

2. Secondary Outcome: Renal Safety Endpoint
Description: Number of patients with doubling of the serum creatinine or plasma cystatin C value compared to baseline with an absolute value >2 mg/dL or >2 mg/L, respectively, or the need for ultrafiltration and/or renal replacement therapy during the index hospital admission.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 52 | 51
Participants | 9 | 3

3. Secondary Outcome: Hemodynamic Safety Endpoint
Description: Number of patients with a ystolic blood pressure <90 mmHg or mean arterial pressure <65 mmHg or need for vasopressors and/or inotropes during the index hospital admission.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 52 | 51
Participants | 10 | 4

4. Secondary Outcome: Natriuretic Peptide Change After 30 Days
Description: Relative NT-proBNP change from baseline to 30 days after randomisation [%].
Time Frame: 30 days
Population: This endpoint could not be assessed in patients who died (n=3 in the intervention arm and n=4 in the control arm). In addition, 1 patient in the intervention arm withdrew consent during follow-up. Vital status could be assessed, but no blood sample was available for this patient. Finally, 5 blood samples were missing in the control group because patients were unable to physically attend the final follow-up visit.
Measure: Mean (Standard Deviation); unit: % of change from baseline
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 48 | 42
% of change from baseline | -37 (64) | -46 (40)

5. Secondary Outcome: Cancer Antigen 125 (CA125) Change After 30 Days
Description: Relative cancer antigen 125 (CA125) change from baseline to 30 days after randomisation [%].
Time Frame: 30 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: % of change from baseline
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 48 | 42
% of change from baseline | -69 (40) | -21 (68)

6. Secondary Outcome: Number of Participants With Successful Clinical Decongestion
Description: Number of participants with no more than trace edema, absence of jugular venous distension and no rales upon the moment of transition from intravenous diuretics to oral diuretic therapy according to the protocol.
Time Frame: 30 days
Population: This endpoint was not be assessed in patients who died (n=3 in the intervention arm and n=4 in the control arm). One edema score was missing in the control group and could not be retrieved, precluding the assessment of decongestion success.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 49 | 46
Participants | 33 | 26

7. Secondary Outcome: Length of Intravenous Diuretic Therapy
Description: Number of consecutive days from randomization during the index admission on which intravenous diuretic therapy was administered.
Time Frame: 30 days
Population: This endpoint was not be assessed in patients who died (n=3 in the intervention arm and n=4 in the control arm).
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 49 | 47
days | 4 [3 to 5] | 4 [3 to 6.5]

8. Secondary Outcome: Overall Well-being After Decongestion
Description: Five-point Likert scale for overall well-being upon the moment of transition from intravenous diuretics to oral diuretic therapy according to the protocol and compared with the moment of randomisation (5: much improved/4: slightly improved/3: neutral/2: slightly worse/1: much worse).
Time Frame: 30 days
Population: This endpoint could not be assessed in patients who died before switching to oral diuretics (n=1 in the intervention group and n=3 in the control group).
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 51 | 48
Participants
  Significantly worse | 0 | 0
  Worse | 3 | 0
  Unchanged | 3 | 4
  Better | 28 | 35
  Significantly better | 17 | 9

9. Secondary Outcome: Length of the Index Hospital Admission
Description: Length of the index hospital admission [days].
Time Frame: 30 days
Population: This endpoint was not be assessed in patients who died (n=3 in the intervention arm and n=4 in the control arm).
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 49 | 47
days | 7 [5 to 9] | 7 [5 to 10]

10. Secondary Outcome: Number of Participants Who Are Death, or Have a Non-elective Hospital Admission or Non-elective Medical Contact
Description: Number of participants who are death, or have a non-elective hospital admission or non-elective medical contact
Time Frame: 30 days
Population: One patient in the intervention arm withdrew consent during follow-up. Vital status could be assessed, but not data on hospitalizations or medical contacts. Therefore the overall number of participants analyzed is 1 lower than for the primary endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Control Arm
Number analyzed (Participants) | 51 | 51
Participants | 9 | 12

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Intervention Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 3/52 | 4/51
Serious Adverse Events (participants affected / at risk) | 6/52 | 14/51
Other Adverse Events (participants affected / at risk) | 13/52 | 21/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=52) | Control Arm (N=51)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 3 (3) — leading to hospital admission or need for renal replacement therapy
Worsening heart failure (Cardiac disorders) | 1 (1) | 7 (7) — administration of intravenous diuretics or intensification of oral diuretics leading to hospital admission or urgent evaluation
Urgent electrical cardioversion of atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Symptomatic bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Hyperkalaemia (Renal and urinary disorders) | 0 (0) | 1 (1) — leading to hospitalization
Hypocalcemia (Endocrine disorders) | 1 (1) | 0 (0) — leading to hospitalization
Need for vasopressor (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Arm (N=52) | Control Arm (N=51)
Hypokalaemia (Renal and urinary disorders) | 13 (13) | 21 (21) — <3.5 mmol/L

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/91/NCT05411991/Prot_003.pdf
  • Statistical Analysis Plan (2024-06-23): https://cdn.clinicaltrials.gov/large-docs/91/NCT05411991/SAP_002.pdf